CLINICAL TRIAL: NCT02293395
Title: A Randomized, Double-Blind, Double-Dummy, Active-controlled, Parallel-group, Multicenter Study to Compare the Safety of Rivaroxaban Versus Acetylsalicylic Acid in Addition to Either Clopidogrel or Ticagrelor Therapy in Subjects With Acute Coronary Syndrome
Brief Title: A Study to Compare the Safety of Rivaroxaban Versus Acetylsalicylic Acid in Addition to Either Clopidogrel or Ticagrelor Therapy in Participants With Acute Coronary Syndrome
Acronym: GEMINI ACS 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bayer (Industry); Duke Clinical Research Institute (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR106261; RIVAROXACS2002 (Other: Janssen Research & Development, LLC); 2014-004266-26 (EudraCT Number)
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Myocardial infarction; Unstable angina; Acetylsalicylic acid; Rivaroxaban; JNJ-39039039; Bay 59-7939; Xarelto; Clopidogrel; Ticagrelor; Plavix; Brilinta; Effient
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable | interventions — Aspirin; Rivaroxaban; Clopidogrel; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (4):
- Stratum 1/ASA (Active Comparator): Acetylsalicylic acid (ASA) 100 milligram (mg) enteric-coated tablet once daily orally along with clopidogrel 75 mg once daily orally, up to either 180 days after randomization of the last enrolled participant in the study or Day 360, whichever occurs earlier.
  Interventions: Drug: Acetylsalicylic acid; Drug: Clopidogrel
- Stratum 1/Rivaroxaban (Experimental): Rivaroxaban 2.5 mg tablet twice daily orally along with clopidogrel 75 mg once daily orally, up to either 180 days after randomization of the last enrolled participant in the study or Day 360, whichever occurs earlier.
  Interventions: Drug: Rivaroxaban; Drug: Clopidogrel
- Stratum 2/ASA (Active Comparator): ASA 100 mg enteric-coated tablet once daily orally along with ticagrelor 90 mg twice daily orally, up to either 180 days after randomization of the last enrolled participant in the study or Day 360, whichever occurs earlier.
  Interventions: Drug: Acetylsalicylic acid; Drug: Ticagrelor
- Stratum 2/Rivaroxaban (Experimental): Rivaroxaban 2.5 mg tablet twice daily orally along with ticagrelor 90 mg twice daily orally, up to either 180 days after randomization of the last enrolled participant in the study or Day 360, whichever occurs earlier.
  Interventions: Drug: Rivaroxaban; Drug: Ticagrelor

INTERVENTIONS:
Drug: Acetylsalicylic acid — ASA 100 mg enteric-coated tablet once daily orally.
  Other Names: Aspirin
  Arms: Stratum 1/ASA; Stratum 2/ASA
Drug: Rivaroxaban — Rivaroxaban 2.5 mg tablet twice daily orally.
  Other Names: JNJ-39039039; Bay 59-7939; Xarelto
  Arms: Stratum 1/Rivaroxaban; Stratum 2/Rivaroxaban
Drug: Clopidogrel — Clopidogrel 75 mg once daily orally.
  Other Names: Plavix
  Arms: Stratum 1/ASA; Stratum 1/Rivaroxaban
Drug: Ticagrelor — Ticagrelor 90 mg twice daily orally.
  Other Names: Brilinta
  Arms: Stratum 2/ASA; Stratum 2/Rivaroxaban

SUMMARY:
The purpose of this study is to estimate the risk of bleeding with rivaroxaban, compared with acetylsalicylic acid (ASA), in addition to a single antiplatelet/ platelet adenosine diphosphate P2Y12 receptor antagonist (P2Y12 inhibitor agent: clopidogrel or ticagrelor), in participants with a recent acute coronary syndrome (ACS: including ST segment elevation myocardial infarction [STEMI] and non-ST-segment elevation acute coronary syndrome [NSTE-ACS]).

DETAILED DESCRIPTION:
This is a prospective, randomized (the study drug is assigned by chance), double-blind (neither physician nor participant knows the treatment that the participant receives), active-controlled (study in which the experimental treatment or procedure is compared to a standard treatment or procedure), parallel group (each group of participants will be treated at the same time), multicenter (when more than one hospital or medical school team work on a medical research study) study in participants with a recent ACS (STEMI or NSTE-ACS). All the eligible participants receiving background treatment of ASA plus clopidogrel (Stratum 1) or ASA plus ticagrelor (Stratum 2) will be randomly assigned to either receive ASA or rivaroxaban on background of P2Y12 receptor antagonists treatment. This study will include 3 phases: Screening Phase (up to 10 days, before study start on Day 1), Double-blind Treatment Phase (up to either 180 days after randomization of the last enrolled participant in the study or Day 360, whichever occurs earlier), and Follow-up Phase (up to 30 days). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants, 18 years or older, must have symptoms suggestive of acute coronary syndrome (ACS) (angina, or symptoms thought to be equivalent) within 48 hours of hospital presentation, or developed ACS while being hospitalized, and has a diagnosis of: a) ST segment elevation myocardial infarction (STEMI); b) non-ST-segment elevation acute coronary syndrome (NSTE-ACS). However, participant who is 54 years of age or younger must also have either diabetes mellitus or a history of a prior myocardial infarction (MI), in addition to the presenting ACS event
* Participant must be randomized within the screening window of 10 days after hospital admission for the index ACS event. Participant should have received acute phase treatment for the index ACS, such as intravenous anticoagulant or antiplatelet, and are receiving maintenance dual antiplatelet therapy (DAPT) with either clopidogrel plus acetyl salicylic acid (ASA), or ticagrelor plus ASA, with the intent to continue the treatment with a platelet adenosine diphosphate P2Y12 receptor antagonist (P2Y12 inhibitor) after randomization
* Participants must agree to provide a pharmacogenomics deoxyribonucleic acid (DNA) sample

Exclusion Criteria:

* Participant has any conditions that, in the opinion of the investigator, contraindicates anticoagulant therapy or would have an unacceptable risk
* Participant with a prior stroke of any etiology or transient ischemic attack (TIA)
* Participant who received thrombolytic therapy as treatment for the index ACS event cannot be enrolled in the ticagrelor stratum
* Participant has anticipated need for chronic administration of omeprazole or esomeprazole concomitantly with clopidogrel
* Participant has known allergy or intolerance to ASA or rivaroxaban

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3037 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (259):
- United States (49):
  - Alexander City, Alabama
  - Banning, California
  - Sylmar, California
  - Aurora, Colorado
  - Littleton, Colorado
  - Jupiter, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Athens, Georgia
  - Cumming, Georgia
  - Macon, Georgia
  - Tucker, Georgia
  - Boise, Idaho
  - Coeur d'Alene, Idaho
  - Jerseyville, Illinois
  - Indianapolis, Indiana
  - Munster, Indiana
  - Bay City, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Mount Clemens, Michigan
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - St Louis, Missouri
  - Kalispell, Montana
  - Stony Brook, New York
  - Rocky Mount, North Carolina
  - Sanford, North Carolina
  - Cincinnati, Ohio
  - Zanesville, Ohio
  - Bartlesville, Oklahoma
  - Tulsa, Oklahoma
  - Abington, Pennsylvania
  - Langhorne, Pennsylvania
  - Philadelphia, Pennsylvania
  - Sayre, Pennsylvania
  - York, Pennsylvania
  - Rapid City, South Dakota
  - Oak Ridge, Tennessee
  - Amarillo, Texas
  - Fort Sam Houston, Texas
  - Houston, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Danville, Virginia
  - Puyallup, Washington
- Argentina (13):
  - Buenos Aires
  - Caba
  - Ciudad de Buenos Aires
  - Cordooba
  - Corrientes
  - Córdoba
  - La Plata
  - Mar del Plata
  - Resistencia
  - Rosario
  - Salta
  - San Martín
  - Santa Fe
- Australia (11):
  - Brisbane
  - Cairns
  - Chermside
  - Elizabeth Vale
  - Herston
  - Hobart
  - Launceston
  - Liverpool
  - Murdoch
  - Nambour
  - New Lambton Heights
- Belgium (13):
  - Antwerp
  - Bonheiden
  - Brasschaat
  - Bruges
  - Edegem
  - Genk
  - Ghent
  - Huy
  - Liège
  - Mol
  - Roeselare
  - Ronse
  - Turnhout
- Brazil (15):
  - Belo Horizonte
  - Blumenau
  - Campina Grande do Sul
  - Campinas
  - Curitiba
  - Marília
  - Passo Fundo
  - Porto Alegre
  - Recife
  - Salvador
  - São José do Rio Preto
  - São Paulo
  - Tatuí
  - Uberlândia
  - Votuporanga
- Bulgaria (10):
  - Blagoevgrad
  - Burgas
  - Haskovo
  - Lovech
  - Pazardzhik
  - Pleven
  - Rousse
  - Sandanski
  - Sofia
  - Varna
- Canada (11):
  - Edmonton, Alberta
  - New West Minister, British Columbia
  - Victoria, British Columbia
  - Greater Sudbury, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saint-Charles-Borromée, Quebec
  - Sherbrooke, Quebec
  - Québec
- Czechia (7):
  - Brno
  - Kolin Iii.
  - Ostrava
  - Plzen-Bory
  - Prague
  - Třebíč
  - Znojmo
- Denmark (3):
  - Herlev
  - Køge
  - Silkeborg
- France (8):
  - Besançon
  - Chambray-lès-Tours
  - Jossigny
  - Le Coudray
  - Lyon
  - Montauban
  - Nantes
  - Périgueux
- Hungary (10):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Győr
  - Gyula
  - Kaposvár
  - Kecskemét
  - Nyíregyháza
  - Székesfehérvár
  - Szolnok
- Japan (14):
  - Gifu
  - Kagawa
  - Kitakyushu
  - Kobe
  - Kumamoto
  - Matsue
  - Nagano
  - Osaka
  - Sayama-Shi
  - Tokyo
  - Uwajima-Shi
  - Yokohama
  - Yonago
  - Yotsui 2-8-1
- Netherlands (13):
  - 's-Hertogenbosch
  - Amersfoort
  - Amsterdam
  - Blaricum
  - Den Helder
  - Gouda
  - Groningen
  - Hoofddorp
  - Hoogeveen
  - Nijmegen
  - Rotterdam
  - Schiedam
  - The Hague
- Poland (20):
  - Bielsko-Biala
  - Bytom
  - Chrzanów
  - Dąbrowa Górnicza
  - Gdynia
  - Grodzisk Mazowiecki
  - Inowrocław
  - Kędzierzyn-Koźle
  - Kielce
  - Koszalin
  - Krakow
  - Lodz
  - Nowy Targ
  - Nysa
  - Oświęcim
  - Polanica-Zdrój
  - Puławy
  - Tychy
  - Warsaw
  - Włocławek
- Russia (18):
  - Barnaul
  - Chita
  - Ivanovo
  - Kaliningrad
  - Kemerovo
  - Krasnodar
  - Krasnoyarsk
  - Moscow
  - Nizhny Novgorod
  - Orenburg
  - Penza
  - Perm
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Syktyvkar
  - Tyumen
  - Yekaterinburg
- South Korea (5):
  - Gwangju
  - Incheon
  - Seongnam
  - Seoul
  - Suwon
- Spain (9):
  - A Coruña
  - Almería
  - Ávila
  - Barcelona
  - Madrid
  - Málaga
  - Murcia
  - Sant Boi de Llobregat
  - Tarragona
- Sweden (9):
  - Falun
  - Jönköping
  - Linköping
  - Lund
  - Örebro
  - Östersund
  - Stockholm
  - Sundsvall
  - Uppsala
- Turkey (Türkiye) (11):
  - Adana
  - Ankara
  - Aydin
  - Bursa
  - Diyarbakır
  - Eskişehir
  - Istanbul
  - Kahramanmaraş
  - Kocaeli
  - Konya
  - Sivas
- Ukraine (10):
  - Cherkasy
  - Dnipropetrovsk
  - Kharkiv
  - Kyiv
  - Lutsk
  - Lviv
  - Odesa
  - Ternopil
  - Zaporizhzhia
  - Zhytomyr

REFERENCES:
- [Derived] Gibson WJ, Nafee T, Travis R, Yee M, Kerneis M, Ohman M, Gibson CM. Machine learning versus traditional risk stratification methods in acute coronary syndrome: a pooled randomized clinical trial analysis. J Thromb Thrombolysis. 2020 Jan;49(1):1-9. doi: 10.1007/s11239-019-01940-8. PMID 31535314
- [Derived] Povsic TJ, Ohman EM, Roe MT, White J, Rockhold FW, Montalescot G, Cornel JH, Nicolau JC, Steg PG, James S, Bode C, Welsh RC, Plotnikov AN, Mundl H, Gibson CM. P2Y12 Inhibitor Switching in Response to Routine Notification of CYP2C19 Clopidogrel Metabolizer Status Following Acute Coronary Syndromes. JAMA Cardiol. 2019 Jul 1;4(7):680-684. doi: 10.1001/jamacardio.2019.1510. PMID 31141104
- [Derived] Ohman EM, Roe MT, Steg PG, James SK, Povsic TJ, White J, Rockhold F, Plotnikov A, Mundl H, Strony J, Sun X, Husted S, Tendera M, Montalescot G, Bahit MC, Ardissino D, Bueno H, Claeys MJ, Nicolau JC, Cornel JH, Goto S, Kiss RG, Guray U, Park DW, Bode C, Welsh RC, Gibson CM. Clinically significant bleeding with low-dose rivaroxaban versus aspirin, in addition to P2Y12 inhibition, in acute coronary syndromes (GEMINI-ACS-1): a double-blind, multicentre, randomised trial. Lancet. 2017 May 6;389(10081):1799-1808. doi: 10.1016/S0140-6736(17)30751-1. Epub 2017 Mar 18. PMID 28325638
- [Derived] Povsic TJ, Roe MT, Ohman EM, Steg PG, James S, Plotnikov A, Mundl H, Welsh R, Bode C, Gibson CM. A randomized trial to compare the safety of rivaroxaban vs aspirin in addition to either clopidogrel or ticagrelor in acute coronary syndrome: The design of the GEMINI-ACS-1 phase II study. Am Heart J. 2016 Apr;174:120-8. doi: 10.1016/j.ahj.2016.01.004. Epub 2016 Jan 18. PMID 26995378

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 3,145 participants were screened for eligibility, of these 108 participants were screening failures and the remaining 3,037 participants were randomized.
Groups:
- Rivaroxaban 2.5 mg Twice Daily (BID): Participants received oral dose of 2.5 mg rivaroxaban BID and acetylsalicylic acid (ASA) placebo once daily (OD) along with either clopidogrel 75 mg OD or ticagrelor 90 mg BID for a minimum of 180 days, and up to 360 days of treatment.
- Acetylsalicylic Acid 100 mg Once Daily (OD): Participants received oral dose of 100 mg ASA OD and rivaroxaban placebo BID along with either clopidogrel 75 mg OD or ticagrelor 90 mg BID for a minimum of 180 days, and up to 360 days of treatment.
Period: Overall Study
Arm/Group | Rivaroxaban 2.5 mg Twice Daily (BID) | Acetylsalicylic Acid 100 mg Once Daily (OD)
Started | 1519 | 1518
Treated | 1510 | 1506
Completed | 1510 | 1511
Not Completed | 9 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban 2.5 mg Twice Daily (BID) | Acetylsalicylic Acid 100 mg Once Daily (OD) | Total
Number analyzed (Participants) | 1519 | 1518 | 3037
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.14) | 62.9 (8.82) | 62.8 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 385 | 377 | 762
  Male | 1134 | 1141 | 2275
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1417 | 1407 | 2824
  Black | 24 | 16 | 40
  Asian | 54 | 63 | 117
  Others | 24 | 32 | 56
Region of Enrollment [Number; unit: participants]
  ARGENTINA | 66 | 65 | 131
  AUSTRALIA | 18 | 17 | 35
  BELGIUM | 49 | 40 | 89
  BRAZIL | 77 | 85 | 162
  BULGARIA | 83 | 78 | 161
  CANADA | 37 | 47 | 84
  CZECH REPUBLIC | 34 | 37 | 71
  DENMARK | 1 | 2 | 3
  FRANCE | 28 | 29 | 57
  HUNGARY | 101 | 100 | 201
  ITALY | 75 | 59 | 134
  JAPAN | 26 | 33 | 59
  NETHERLANDS | 69 | 65 | 134
  POLAND | 158 | 175 | 333
  RUSSIA | 237 | 244 | 481
  SPAIN | 62 | 60 | 122
  SWEDEN | 42 | 37 | 79
  TURKEY | 102 | 98 | 200
  UKRAINE | 137 | 129 | 266
  UNITED STATES | 93 | 88 | 181
  Korea, Republic Of | 24 | 30 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non Coronary Artery Bypass Graft-Related (Non CABG-related) Thrombolysis in Myocardial Infarction (TIMI) Clinically Significant Bleeding Events
Description: Non CABG-related TIMI clinically significant bleeding events are sum of non CABG-related TIMI major bleeding events, TIMI minor bleeding events and TIMI bleeding events requiring medical attention. Major: any symptomatic intracranial bleeding: clinically overt signs of hemorrhage with hemoglobin (Hb) drop of greater than or equal to (>=)5 gram per deciliter (g/dl) (or absolute drop in hematocrit of >=15%) and fatal bleeding (results in death within 7 days); Minor: clinically overt sign of hemorrhage with Hb drop of 3 - <5 g/dl (or drop in hematocrit of 9 - <15%); requiring medical attention: bleeding event that required medical, surgical treatment/laboratory evaluation and did not meet criteria for major/minor bleeding event.
Time Frame: From start of study treatment until follow-up (up to 390 days)
Population: Population analyzed included all randomized participants who had received at least one dose of study agent and had events that occurred between randomization and the last dose of the study agent plus 2 days or untreated participants who had events that occurred between randomization to 2 days thereafter.
Measure: Number; unit: participants
Arm/Group | Rivaroxaban 2.5 mg Twice Daily (BID) | Acetylsalicylic Acid 100 mg Once Daily (OD)
Number analyzed (Participants) | 1519 | 1518
participants | 80 | 74
Statistical Analysis 1: Comparison: Rivaroxaban 2.5 mg Twice Daily (BID) vs Acetylsalicylic Acid 100 mg Once Daily (OD); Test type: Superiority or Other; p = 0.584, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.8 to 1.5]

ADVERSE EVENTS:
Time Frame: Up to 390 days
Description: Population analyzed included all randomized participants who had received at least one dose of study drug and had events between randomization and last dose of study drug +2 days. No comparison of adverse events between strata was planned.
Arm/Group | Rivaroxaban 2.5 mg Twice Daily (BID) | Acetylsalicylic Acid 100 mg Once Daily (OD)
Serious Adverse Events (participants affected / at risk) | 125/1510 | 138/1506
Other Adverse Events (participants affected / at risk) | 81/1510 | 84/1506
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban 2.5 mg Twice Daily (BID) (N=1510) | Acetylsalicylic Acid 100 mg Once Daily (OD) (N=1506)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute Left Ventricular Failure (Cardiac disorders) | 3 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 2
Angina Unstable (Cardiac disorders) | 5 | 5
Aortic Valve Stenosis (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 3 | 7
Atrial Flutter (Cardiac disorders) | 1 | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 9 | 7
Cardiac Failure Acute (Cardiac disorders) | 1 | 0
Cardiac Failure Chronic (Cardiac disorders) | 3 | 0
Cardiac Failure Congestive (Cardiac disorders) | 2 | 1
Cardiac Ventricular Thrombosis (Cardiac disorders) | 1 | 0
Cardiovascular Insufficiency (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 2 | 0
Coronary Artery Stenosis (Cardiac disorders) | 1 | 1
Intracardiac Thrombus (Cardiac disorders) | 1 | 1
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0
Myocardial Fibrosis (Cardiac disorders) | 0 | 2
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Myocardial Rupture (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Pleuropericarditis (Cardiac disorders) | 1 | 0
Postinfarction Angina (Cardiac disorders) | 0 | 1
Sinus Arrest (Cardiac disorders) | 0 | 1
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Chronic Gastritis (Gastrointestinal disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Diverticulum Intestinal (Gastrointestinal disorders) | 1 | 0
Erosive Oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Pancreatic Necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 2
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 2 | 2
Death (General disorders) | 0 | 1
Implant Site Ulcer (General disorders) | 0 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Stent-Graft Endoleak (General disorders) | 0 | 1
Vascular Stent Restenosis (General disorders) | 1 | 0
Vascular Stent Stenosis (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 3 | 5
Cholelithiasis (Hepatobiliary disorders) | 3 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 1 | 0
H1n1 Influenza (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Infectious Pleural Effusion (Infections and infestations) | 0 | 1
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 0
Orchitis (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 5
Postoperative Wound Infection (Infections and infestations) | 0 | 1
Pyelonephritis Chronic (Infections and infestations) | 2 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Spinal Cord Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 1 | 3
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1
Heat Illness (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 2
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna Fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Site Pain (Injury, poisoning and procedural complications) | 1 | 0
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Cardiac Stress Test Abnormal (Investigations) | 0 | 2
Haemoglobin Decreased (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0
Liver Function Test Increased (Investigations) | 1 | 0
Mediastinoscopy (Investigations) | 1 | 0
Weight Decreased (Investigations) | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Ligamentitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rapidly Progressive Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix Carcinoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary Gland Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vascular Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0
Facial Paralysis (Nervous system disorders) | 0 | 1
Intracranial Aneurysm (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 3
Vertebral Artery Stenosis (Nervous system disorders) | 0 | 1
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 2
Panic Attack (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Nephropathy Toxic (Renal and urinary disorders) | 1 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 0 | 1
Renal Colic (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 2 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Inguinal Hernia Repair (Surgical and medical procedures) | 0 | 1
Lung Neoplasm Surgery (Surgical and medical procedures) | 0 | 1
Lymphadenectomy (Surgical and medical procedures) | 0 | 1
Aortic Aneurysm (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Brachiocephalic Arteriosclerosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive Crisis (Vascular disorders) | 5 | 2
Hypotension (Vascular disorders) | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1
Peripheral Artery Aneurysm (Vascular disorders) | 1 | 0
Peripheral Artery Occlusion (Vascular disorders) | 0 | 1
Peripheral Artery Stenosis (Vascular disorders) | 1 | 1
Subclavian Artery Stenosis (Vascular disorders) | 1 | 0
Vascular Occlusion (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban 2.5 mg Twice Daily (BID) (N=1510) | Acetylsalicylic Acid 100 mg Once Daily (OD) (N=1506)
Chest Pain (General disorders) | 11 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 39
Hypertension (Vascular disorders) | 23 | 22

LIMITATIONS AND CAVEATS:
Study population was homogenous with limited participation of non-Caucasian participants. Randomization was not performed for use of P2Y12 inhibitor; strata comparisons between bleeding and efficacy endpoints are confounded and were not planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.